CLINICAL TRIAL: NCT00761774
Title: An Open-label, Multinational, Multicenter, Follow-up Study to Evaluate the Long-term Safety and Efficacy of Brivaracetam Used at a Flexible Dose up to a Maximum of 200 mg/Day in Subjects Aged 16 Years or Older Suffering From Epilepsy.
Brief Title: An Open-label, Multinational, Multicenter, Follow-up Study to Evaluate the Long-term Safety and Efficacy of Brivaracetam
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N01315; 2008-001433-98 (EudraCT Number)
Expanded Access: NCT03532516 (Available)
Record Dates: First submitted 2008-09-26; First posted 2008-09-30 (Estimated); Results first posted 2018-04-23 (Actual); Last update posted 2018-07-11 (Actual); Status verified 2018-03

CONDITIONS: Epilepsy
Keywords: Epilepsy; Monotherapy; Partial Onset Seizures
MeSH Terms: conditions — Epilepsy | interventions — brivaracetam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Brivaracetam (Experimental): Brivaracetam at flexible dosing up to 200mg /day
  Interventions: Drug: Brivaracetam

INTERVENTIONS:
Drug: Brivaracetam — Subjects will begin at a recommended dose of Brivaracetam 100 mg/day. Subjects will continue treatment at a dose up to a maximum of 200 mg/day with a twice per day administration. Up- and down-titration steps may be performed in steps of a maximum of 50 mg/day on a weekly basis. Full down-titration should include a one week step on 20 mg/day. The study medication will come in 10 mg and 25 mg tablet strengths.
  Other Names: ucb 34714

SUMMARY:
The Sponsor wishes to develop brivaracetam as an anti-epileptic treatment in subjects 16 years and older with epilepsy. This study permits continued access to treatment for subjects who participated in a previous epilepsy study. The study will explore the long-term safety and efficacy of brivaracetam.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with epilepsy who participated in previous brivaracetam trials which allow access to the present trial.
* Subjects from whom the Investigator believes a reasonable potential benefit from the long-term administration of brivaracetam may be expected.

Exclusion Criteria:

• Severe medical, neurological and psychiatric disorders, including current suicidal ideation or behaviour, or laboratory values which may have an impact on the safety of the subject, as determined by the investigator.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2008-11; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — +1 844 599 2273(UCB)
Locations (58):
- United States (25):
  - 304, Phoenix, Arizona
  - 281, Fresno, California
  - 288, Pasadena, California
  - 240, Riverside, California
  - 245, Sacramento, California
  - 285, Peoria, Illinois
  - 224, Indianapolis, Indiana
  - 266, Lexington, Kentucky
  - 231, Waldorf, Maryland
  - 278, Burlington, Massachusetts
  - 270, New York, New York
  - 284, Hickory, North Carolina
  - 241, Columbus, Ohio
  - 265, Oklahoma City, Oklahoma
  - 297, Germantown, Tennessee
  - 260, Austin, Texas
  - 236, Bedford, Texas
  - 267, Dallas, Texas
  - 268, Houston, Texas
  - 211, Layton, Utah
  - 235, Ogden, Utah
  - 218, Burlington, Vermont
  - 279, Danville, Virginia
  - 277, Charleston, West Virginia
  - 213, Marshfield, Wisconsin
- Australia (4):
  - 400, Chatswood, New South Wales
  - 404, Adelaide, South Australia
  - 402, Fitzroy, Victoria
  - 401, Parkville, Victoria
- Belgium (2):
  - 004, Ghent
  - 003, Kortrijk
- Canada (3):
  - 205, Calgary, Alberta
  - 203, Edmonton, Alberta
  - 206, Toronto, Ontario
- Czechia (5):
  - 023, Brno
  - 020, Litomyšl
  - 021, Ostava
  - 024, Ostrava-Trebovice
  - 026, Prague
- France (2):
  - 040, Béthune
  - 041, Toulouse
- Germany (6):
  - 055, Berlin
  - 056, Bernau
  - 054, Bielefeld
  - 063, Mainz
  - 051, München
  - 065, Regensburg
- Hungary (2):
  - 072, Budapest
  - 074, Budapest
- Italy (5):
  - 084, Bergamo
  - 082, Messina
  - 085, Orbassano
  - 083, Perugia
  - 080, Pisa
- 090, Madrid, Spain
- Sweden (3):
  - 100, Gothenburg
  - 102, Lund
  - 101, Stockholm

REFERENCES:
- [Derived] Markham A. Brivaracetam: First Global Approval. Drugs. 2016 Mar;76(4):517-22. doi: 10.1007/s40265-016-0555-6. PMID 26899665
- See also: Product Information — https://www.briviact.com/briviact-PI.pdf?v=1479491757
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll patients in November 2008 and concluded in March 2017.
Pre-assignment Details: Participant Flow refers to the Safety Set, which consisted of all subjects who took at least 1 dose of study drug.
Groups:
- Brivaracetam: This arm consisted of subjects who received Brivaracetam (BRV) at flexible dosing up to 200 mg/day.
Period: Overall Study
Arm/Group | Brivaracetam
Started | 108
Completed | 29
Not Completed | 79
Not completed — Adverse Event | 17
Not completed — Lack of Efficacy | 37
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 9
Not completed — Non-compliance | 4
Not completed — End of study | 2
Not completed — Reclassification of seizures | 1
Not completed — Medical decision to read SUSAR reports | 1
Not completed — Sponsor decision | 1
Not completed — Investigator clinical judgement | 1
Not completed — Patient moved out of study area | 1
Not completed — Coordinator leaving site | 1
Not completed — Subject IP non-compliance | 1
Not completed — IP stopped by hospital physician | 1

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to the Safety Set which consisted of all subjects who received at least 1 dose of study medication.
Arm/Group | Brivaracetam
Number analyzed (Participants) | 108
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 103
  >=65 years | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.8 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56
  Male | 52
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 7
  White | 97
  Other/Mixed | 4

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With at Least One Treatment-emergent Adverse Event (TEAE) During the Evaluation Period From Entry Visit 1 Through End of Treatment (up to 9 Years)
Description: Treatment-emergent Adverse events (TEAE) are any untoward medical occurrences in a subject during administered study treatment, whether or not these events are related to study treatment.
Time Frame: During the Evaluation Period (up to 9 years)
Population: The Safety Analysis Set consisted of all subjects who took at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Groups:
- Brivaracetam (SS): This arm consisted of subjects who received Brivaracetam (BRV) at flexible dosing up to 200 mg/day.
Arm/Group | Brivaracetam (SS)
Number analyzed (Participants) | 108
percentage of participants | 90.7

2. Primary Outcome: Percentage of Subjects Who Withdrew Due to Adverse Event (AE) During the Evaluation Period From Entry Visit 1 Through End of Treatment (up to 9 Years)
Description: Adverse Events (AE) are any untoward medical occurrences in a subject during administered study treatment, whether or not these events are related to study treatment.
Time Frame: During the Evaluation Period (up to 9 years)
Population: The Safety Analysis Set consisted of all subjects who took at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Groups:
- Brivaracetam (SS): This arm consisted of subjects who received Brivaracetam (BRV) at flexible dosing up to 200mg/day.
Arm/Group | Brivaracetam (SS)
Number analyzed (Participants) | 108
percentage of participants | 15.7

3. Primary Outcome: Percentage of Subjects With a Serious Adverse Event (SAE) During the Evaluation Period From Entry Visit 1 Through End of Treatment (up to 9 Years)
Description: An SAE was any untoward medical occurrence that, at any dose resulted in death, was life threatening, required in-subject hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, or was a congenital anomaly/birth defect.
Time Frame: During the Evaluation Period (up to 9 years)
Population: The Safety Analysis Set consisted of all subjects who took at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Brivaracetam (SS)
Number analyzed (Participants) | 108
percentage of participants | 24.1

4. Secondary Outcome: Percentage of Subjects on Continuous Brivaracetam Monotherapy for at Least 3 Months of the Evaluation Period (up to 9 Years)
Description: BRV monotherapy is defined as continuous treatment with BRV only (ie, no treatment with another anti-epileptic drug (AED)). Use of rescue AED for a duration of no more than 2 consecutive days will not disqualify a subject from being defined as on continuous monotherapy provided the use of rescue AED does not exceed more than 1 time per week.
Time Frame: During the Evaluation Period (up to 9 years)
Population: The Efficacy Analysis Set consisted of all subjects who took at least 1 dose of study drug and had at least 1 seizure Daily Record Card (DRC) day during the Evaluation Period.
Measure: Number; unit: percentage of participants
Groups:
- Brivaracetam (ES): This arm consisted of subjects who received Brivaracetam (BRV) at flexible dosing up to 200 mg/day.
Arm/Group | Brivaracetam (ES)
Number analyzed (Participants) | 108
percentage of participants | 38.89

5. Secondary Outcome: Percentage of Subjects on Continuous Brivaracetam Monotherapy for at Least 6 Months, of the Evaluation Period (up to 9 Years)
Description: as for outcome 4
Time Frame: During the Evaluation Period (up to 9 years)
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Brivaracetam (ES)
Number analyzed (Participants) | 108
percentage of participants | 32.41

6. Secondary Outcome: Percentage of Subjects on Continuous Brivaracetam Monotherapy for at Least 12 Months of the Evaluation Period (up to 9 Years)
Description: as for outcome 4
Time Frame: During the Evaluation Period (up to 9 years)
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Brivaracetam (ES)
Number analyzed (Participants) | 108
percentage of participants | 25

ADVERSE EVENTS:
Time Frame: Adverse events were collected throughout the study (up to 9 years).
Arm/Group | Brivaracetam (SS)
All-Cause Mortality (participants affected / at risk) | 1/108
Serious Adverse Events (participants affected / at risk) | 26/108
Other Adverse Events (participants affected / at risk) | 81/108
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Brivaracetam (SS) (N=108)
Angina pectoris (Cardiac disorders) | 3 (3)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Cardiac failure congestive (Cardiac disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Sudden unexplained death in epilepsy (General disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 2 (2)
Pneumonia (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 2 (3)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1)
Intentional overdose (Injury, poisoning and procedural complications) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (1)
Snake bite (Injury, poisoning and procedural complications) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Convulsion (Nervous system disorders) | 5 (7)
Dysarthria (Nervous system disorders) | 1 (1)
Epilepsy (Nervous system disorders) | 1 (1)
Grand mal convulsion (Nervous system disorders) | 2 (4)
Hemiparesis (Nervous system disorders) | 1 (1)
Migraine (Nervous system disorders) | 1 (1)
Monoplegia (Nervous system disorders) | 1 (1)
Postictal state (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Factitious disorder (Psychiatric disorders) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 1 (2)
Somnambulism (Psychiatric disorders) | 1 (2)
Suicide attempt (Psychiatric disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pregnancy of partner (Social circumstances) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Brivaracetam (SS) (N=108)
Diarrhoea (Gastrointestinal disorders) | 12 (16)
Abdominal pain (Gastrointestinal disorders) | 9 (12)
Nausea (Gastrointestinal disorders) | 9 (11)
Toothache (Gastrointestinal disorders) | 7 (10)
Vomiting (Gastrointestinal disorders) | 6 (9)
Fatigue (General disorders) | 17 (19)
Chest pain (General disorders) | 9 (10)
Oedema peripheral (General disorders) | 6 (7)
Nasopharyngitis (Infections and infestations) | 19 (42)
Bronchitis (Infections and infestations) | 8 (13)
Upper respiratory tract infection (Infections and infestations) | 8 (11)
Viral infection (Infections and infestations) | 6 (8)
Fall (Injury, poisoning and procedural complications) | 15 (19)
Contusion (Injury, poisoning and procedural complications) | 9 (11)
Weight increased (Investigations) | 6 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 12 (12)
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 (16)
Convulsion (Nervous system disorders) | 17 (28)
Headache (Nervous system disorders) | 15 (20)
Dizziness (Nervous system disorders) | 14 (18)
Migraine (Nervous system disorders) | 7 (11)
Paraesthesia (Nervous system disorders) | 6 (6)
Tremor (Nervous system disorders) | 6 (7)
Depression (Psychiatric disorders) | 18 (21)
Anxiety (Psychiatric disorders) | 15 (24)
Insomnia (Psychiatric disorders) | 15 (16)
Suicidal ideation (Psychiatric disorders) | 6 (7)
Rash (Skin and subcutaneous tissue disorders) | 13 (16)
Hypertension (Vascular disorders) | 6 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2015-03-25): https://cdn.clinicaltrials.gov/large-docs/74/NCT00761774/Prot_000.pdf
  • Statistical Analysis Plan (2016-06-24): https://cdn.clinicaltrials.gov/large-docs/74/NCT00761774/SAP_001.pdf